CLINICAL TRIAL: NCT06257849
Title: Validity and Reliability of a Danish Version of the Banff Patella Instability Instrument (BPII 2.0-DK)
Status: Active, not recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, PhD, MD, Aarhus University Hospital
Other Study IDs: Questionnaire BPII 2.0-DK
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Patella Dysplasia
Keywords: BPII 2.0; Patella instability; Knee; Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: BPII 2.0 — Banff Patella Instability Instrument 2.0 is a questionnaire developed for measuring outcome in patients with patella instability
  Other Names: Banff Patella Instability Instrument 2.0

SUMMARY:
The Banff Patella Instability Instrument (BPII 2.0) is a disease-specific quality of life questionnaire designed to assess adults with patellar dislocations.

As the BPII 2.0 already is cross-cultural translate and adapted to Danish the examination of the the psychometric properties of the Danish version is still needed

The aim om this study is to determine validity and reliability of the Danish version BPII 2.0-DK in a Danish populations of patients with patellar dislocation.

ELIGIBILITY:
Inclusion Criteria:

* Danish Speaking
* Patella instability problems

Exclusion Criteria:

* None

Ages: 14 Years to 40 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with Patella instability
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Banff patella instability instrument (BPII 2.0) | Baseline, after 6-8 days
  Questionnaire. (0-100 (0 = Worst, 100 = Best))
Anterior knee pain scale (Kujala) | Baseline
  Questionnaire. (0-100 (0 = Worst, 100 = Best))
Victorian Institute of Sports Assessment - Patella questionnaire (VISA-P) | Baseline
  Questionnaire. (0-100 (0 = Worst, 100 = Best))
International knee documentation committee (IKDC) | Baseline
  Questionnaire. (0-100 (0 = Worst, 100 = Best))

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Division of Sports Trauma, Palle Juul-Jensens Boulevard 99, Aarhus N